CLINICAL TRIAL: NCT01774084
Title: Insulin Sensitivity and Beta Cell Function After Carbohydrate Loading in Hip Replacement Surgery: A Randomised Doubled-blinded Control Study
Brief Title: Insulin Sensitivity and Beta Cell Function After Carbohydrate Loading in Hip Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Nystrom, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/3:6
Record Dates: First submitted 2013-01-20; First posted 2013-01-23 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Insulin Sensitivity
Keywords: Insulin sensitivity; Beta cell function; Carbohydrate preload; Elective hip replacement; Double-blind randomized control study
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PreOp, NutriciaNordica AB (Active Comparator): PreOp: 50 kcal/100 mL in the form of maltodextrin and fructose. One bottle of 800 ml to be ingested at bedtime, and at midnight by the latest, and another bottle with 400 ml approximately 2 hours before surgery started.
  Interventions: Dietary Supplement: Experimental: PreOp, NutriciaNordica AB
- Water (Placebo Comparator): Water: One bottle of 800 ml to be ingested at bedtime, and at midnight by the latest, and another bottle with 400 ml approximately 2 hours before surgery started.
  Interventions: Dietary Supplement: Placebo Comparator: Water

INTERVENTIONS:
Dietary Supplement: Experimental: PreOp, NutriciaNordica AB
  Other Names: PreOp, serial number 27 62 95, NutriciaNordica AB
  Arms: PreOp, NutriciaNordica AB
Dietary Supplement: Placebo Comparator: Water
  Arms: Water

SUMMARY:
The purpose of this study is to determine whether preload of carbohydrate or water before elective hip replacement improve insulin sensitivity and or beta cell function in human.

ELIGIBILITY:
Inclusion Criteria:

* Elective hip replacement

Exclusion Criteria:

* Known diabetes mellitus
* Kidney failure (creatinine clearance <40 ml/min
* Liver failure (aspartate and alanine aminotransferases x 2 above reference)
* Hb <110 g/l
* Ongoing severe bacterial or viral infection
* Malignancies
* Psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nyström, MD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Södersjukhuset AB, Stockholm, Sweden
  - Södertälje hospital, Södertälje, Södertälje

REFERENCES:
- [Derived] Ljunggren S, Hahn RG, Nystrom T. Insulin sensitivity and beta-cell function after carbohydrate oral loading in hip replacement surgery: a double-blind, randomised controlled clinical trial. Clin Nutr. 2014 Jun;33(3):392-8. doi: 10.1016/j.clnu.2013.08.003. Epub 2013 Aug 15. PMID 24007934
- See also: Related Info — http://www-ncbi-nlm-nih-gov.proxy.kib.ki.se/pubmed/24007934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitments between December 2011 and November 2012, at Södersjukhuset, Karlolinska Institutet, Stockholm.
Pre-assignment Details: No significant events took part in current studies.
Period: Overall Study
Arm/Group | PreOp, NutriciaNordica AB | Water
Started | 11 | 12
Completed | 10 | 12
Not Completed | 1 | 0
Not completed — Personal reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PreOp, NutriciaNordica AB | Water | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (4) | 68 (4) | 67 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity
Description: Insulin sensitivity is measured by euglycemic hyperinsulinemic clamp
Time Frame: Morning before surgery and up to two days after surgery
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mg/(kg min)
Arm/Group | PreOp, NutriciaNordica AB | Water
Number analyzed (Participants) | 10 | 12
mg/(kg min) | 3.2 (2.8) | 2.4 (2.6)

2. Secondary Outcome: Change in Beta Cell Function
Description: Beta cell function is measured with intravenous glucose tolerance test (IVGTT)
Time Frame: Morning before surgery and up to two days after surgery
Measure: Mean (Standard Deviation); unit: Insulin AUC nmol * min/L
Arm/Group | PreOp, NutriciaNordica AB | Water
Number analyzed (Participants) | 10 | 12
Insulin AUC nmol * min/L | 3.3 (2.4) [2.3 to 3.3] | 2.6 (2.2) [1.7 to 6.4]

ADVERSE EVENTS:
Arm/Group | PreOp, NutriciaNordica AB | Water
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes